CLINICAL TRIAL: NCT05271695
Title: Effect of Dietary Inflammatory Index on Inflammatory Markers and Metabolic Parameters, in Patients With Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Fulya Calikoglu, MD, PhD; Academician; Principle Investigator, Istanbul University
Other Study IDs: 2019/732
Record Dates: First submitted 2022-02-17; First posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Type 2 Diabetes; Dietary Inflammatory Index (DII); Inflammation; Medical Nutrition Therapy
Keywords: Dietary inflammatory index (DII); Inflammation; Type 2 diabetes; inflammatory markers; biochemical parameters
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The patients with type 2 diabetes: * Patients with a diagnosis of Type 2 Diabetes Mellitus and HbA1c ≤ 7%
  * Patients using or not using oral antidiabetic drugs
  * Patients who inject insulin once or twice a day or repeated insulin injections
- The healthy controls: * Patients diagnosed with Type I Diabetes Mellitus,
  * Patients with HbA1c > 7%
  * Those with gestational diabetes,
  * Breastfeeding diabetics,
  * Patients with renal dysfunction,
  * Patients with acute and chronic infection status

SUMMARY:
Nutrition is essential in the treatment and management of Type 2 Diabetes. The importance of adding foods with anti-inflammatory effects to daily diet plans in ensuring glycemic control, preventing the progression of diabetes, and reducing the risk of complications in the future is revealed by new studies added to the literature every day. This study aimed to determine the effects of the dietary inflammatory index (DII) on inflammation markers and metabolic parameters by determining the food consumption status of adults with type 2 diabetes who have good glycemic control.

DETAILED DESCRIPTION:
Nutrition is one of the most important determinants of inflammation. When the results of the studies were examined, it was seen that the diet was associated with inflammation in chronic diseases. It was observed that the consumption of foods such as simple carbohydrates, red meat, saturated fat, and trans fat was associated with high Interleukin-6 (IL-6) levels, which had a pro-inflammatory effect. It has been observed that the consumption of foods such as green leaves, vegetables, fruits, olive oil, whole grains, and fish in the Mediterranean type diet is associated with low levels of inflammation with anti-inflammatory effects. It is known that anti-inflammatory dietary components are essential in preventing chronic diseases. "Diet Inflammatory Index (DII)" was developed to determine the inflammatory load of diets. DII, nutritional components, pro-inflammatory markers C-reactive protein (CRP), Tumor Necrosis Factor Alpha (TNF-α), Interleukin 1 beta (IL-1β) and Interleukin 6 (IL-6) and anti-inflammatory markers Interleukin 10 (IL) -10) is an index provided by evaluating its effect on Interleukin 4 (IL-4). In order to obtain the inflammatory load of the diet, the impact of 45 nutritional parameters on inflammation is calculated. It is calculated as a positive score if the nutrient in the diet has a pro-inflammatory (increasing inflammation) effect and a negative score if it has an anti-inflammatory (reducing inflammation) effect.

Studies conducted with diabetes and DII have observed that feeding individuals with a pro-inflammatory diet cause them to have higher DII scores, higher HbA1c, and an increased risk of developing diabetes.

The primary purpose of this study is to find the relationship between the dietary inflammatory index and inflammatory markers in adult type 2 diabetes patients and to determine whether DII is a valid index in adult type 2 diabetes patients.

The second aim is to evaluate the relationship between DII scores and metabolic parameters in adult type 2 diabetes patients.

With the possible results, it aims to determine the measures to be taken to reduce the chronic inflammatory response due to nutritional status in type 2 diabetes patients and prevent the occurrence of diabetes-related complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of Type 2 Diabetes Mellitus and HbA1c ≤ 7%
* Patients using or not using oral antidiabetic drugs
* Patients who inject insulin once or twice a day or repeated insulin injections

Exclusion Criteria:

* Patients diagnosed with Type I Diabetes Mellitus,
* Patients with HbA1c > 7%
* Those with gestational diabetes,
* Breastfeeding diabetics,
* Patients with renal dysfunction,
* Patients with acute and chronic infection status

Ages: 30 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study was selected among adult type 2 diabetes patients under control at Istanbul University Istanbul Medical Faculty Diabetes Polyclinic between November 2019 and April 2020. The 120 patients included studying were between the ages of 30-74 and were sent to the diet polyclinic by their physicians. As the control group, 30 healthy people from the same age group were included. The data were collected by the researcher by face-to-face interview.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Current serum TNF-α value | At the end of the 10-hour fasting of the patients, a single time
  Serum TNF-α values in the current nutritional status of patients with and without type 2 diabetes will be examined.
Current serum IL-6 value | At the end of the 10-hour fasting of the patients, a single time
  Serum IL-6values in the current nutritional status of patients with and without type 2 diabetes will be examined.
Current serum IL-1β value | At the end of the 10-hour fasting of the patients, a single time
  Serum IL-1β values in the current nutritional status of patients with and without type 2 diabetes will be examined.
Current Dietary Inflammatory Index score | At the end of the 10-hour fasting of the patients, a single time
  The Dietary Inflammatory Index score of the current nutritional status of patients with and without type 2 diabetes will be evaluated. In this study, 31 foods and nutrients were determined from food consumption records. The amounts of nutrients were calculated using the nutrient analysis program. Dietary inflammatory index (DII) score was calculated from these foods.
  In order to calculate the diet inflammatory index score, the z-score must first be calculated. To calculate the Z-score, the standard global consumption amount is subtracted from the average consumption amount of the individual. The result obtained is divided by the standard deviation value. The z score found with this result is converted to the percentile score. The percentile value is multiplied by the full inflammatory effect score. DII is obtained as a result of summing the scores calculated for all nutrients and nutrients. Found DII is an indicator of the inflammatory load of the individual's daily diet.

SECONDARY OUTCOMES:
Current serum glucose value | At the end of the 10-hour fasting of the patients, a single time
Current serum HbA1c value | At the end of the 10-hour fasting of the patients, a single time
Current waist circumference measurement | At the end of the 10-hour fasting of the patients, a single time
Current weight | At the end of the 10-hour fasting of the patients, a single time
Current BMI | At the end of the 10-hour fasting of the patients, a single time
Current fat mass rate | At the end of the 10-hour fasting of the patients, a single time
Current serum HDL value | At the end of the 10-hour fasting of the patients, a single time
Current serum LDL value | At the end of the 10-hour fasting of the patients, a single time
Current serum triglyceride value | At the end of the 10-hour fasting of the patients, a single time
Current serum AST(aspartate aminotransferase) value | At the end of the 10-hour fasting of the patients, a single time
Current serum urea value | At the end of the 10-hour fasting of the patients, a single time
Current serum creatinin value | At the end of the 10-hour fasting of the patients, a single time
Current serum uric acid value | At the end of the 10-hour fasting of the patients, a single time

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Faculty of Medicine, Department of Endocrinology and Metabolism, Istanbul, Capa, Turkey (Türkiye)

REFERENCES:
- [Background] Steckhan N, Hohmann CD, Kessler C, Dobos G, Michalsen A, Cramer H. Effects of different dietary approaches on inflammatory markers in patients with metabolic syndrome: A systematic review and meta-analysis. Nutrition. 2016 Mar;32(3):338-48. doi: 10.1016/j.nut.2015.09.010. Epub 2015 Oct 28. PMID 26706026
- [Background] Cavicchia PP, Steck SE, Hurley TG, Hussey JR, Ma Y, Ockene IS, Hebert JR. A new dietary inflammatory index predicts interval changes in serum high-sensitivity C-reactive protein. J Nutr. 2009 Dec;139(12):2365-72. doi: 10.3945/jn.109.114025. Epub 2009 Oct 28. PMID 19864399
- [Background] Shivappa N, Steck SE, Hurley TG, Hussey JR, Hebert JR. Designing and developing a literature-derived, population-based dietary inflammatory index. Public Health Nutr. 2014 Aug;17(8):1689-96. doi: 10.1017/S1368980013002115. Epub 2013 Aug 14. PMID 23941862
- [Background] Wirth MD, Shivappa N, Steck SE, Hurley TG, Hebert JR. The dietary inflammatory index is associated with colorectal cancer in the National Institutes of Health-American Association of Retired Persons Diet and Health Study. Br J Nutr. 2015 Jun 14;113(11):1819-27. doi: 10.1017/S000711451500104X. Epub 2015 Apr 14. PMID 25871645
- [Background] McGeoghegan L, Muirhead CR, Almoosawi S. Association between an anti-inflammatory and anti-oxidant dietary pattern and diabetes in British adults: results from the national diet and nutrition survey rolling programme years 1-4. Int J Food Sci Nutr. 2015 Aug;67(5):553-61. doi: 10.1080/09637486.2016.1179268. Epub 2016 May 4. PMID 27144647
- [Background] King DE, Xiang J. The Dietary Inflammatory Index Is Associated With Diabetes Severity. J Am Board Fam Med. 2019 Nov-Dec;32(6):801-806. doi: 10.3122/jabfm.2019.06.190092. PMID 31704748
- [Background] Schwingshackl L, Chaimani A, Hoffmann G, Schwedhelm C, Boeing H. A network meta-analysis on the comparative efficacy of different dietary approaches on glycaemic control in patients with type 2 diabetes mellitus. Eur J Epidemiol. 2018 Feb;33(2):157-170. doi: 10.1007/s10654-017-0352-x. Epub 2018 Jan 4. PMID 29302846
- [Background] Benson G, Hayes J. An Update on the Mediterranean, Vegetarian, and DASH Eating Patterns in People With Type 2 Diabetes. Diabetes Spectr. 2020 May;33(2):125-132. doi: 10.2337/ds19-0073. PMID 32425449
- [Background] Meng Y, Bai H, Wang S, Li Z, Wang Q, Chen L. Efficacy of low carbohydrate diet for type 2 diabetes mellitus management: A systematic review and meta-analysis of randomized controlled trials. Diabetes Res Clin Pract. 2017 Sep;131:124-131. doi: 10.1016/j.diabres.2017.07.006. Epub 2017 Jul 8. PMID 28750216
- [Background] Kirkpatrick CF, Bolick JP, Kris-Etherton PM, Sikand G, Aspry KE, Soffer DE, Willard KE, Maki KC. Review of current evidence and clinical recommendations on the effects of low-carbohydrate and very-low-carbohydrate (including ketogenic) diets for the management of body weight and other cardiometabolic risk factors: A scientific statement from the National Lipid Association Nutrition and Lifestyle Task Force. J Clin Lipidol. 2019 Sep-Oct;13(5):689-711.e1. doi: 10.1016/j.jacl.2019.08.003. Epub 2019 Sep 13. PMID 31611148
- [Background] Ley SH, Hamdy O, Mohan V, Hu FB. Prevention and management of type 2 diabetes: dietary components and nutritional strategies. Lancet. 2014 Jun 7;383(9933):1999-2007. doi: 10.1016/S0140-6736(14)60613-9. PMID 24910231
- [Background] Robertson L, Waugh N, Robertson A. Protein restriction for diabetic renal disease. Cochrane Database Syst Rev. 2007 Oct 17;2007(4):CD002181. doi: 10.1002/14651858.CD002181.pub2. PMID 17943769
- [Background] Estruch R, Ros E, Salas-Salvado J, Covas MI, Corella D, Aros F, Gomez-Gracia E, Ruiz-Gutierrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Basora J, Munoz MA, Sorli JV, Martinez JA, Fito M, Gea A, Hernan MA, Martinez-Gonzalez MA; PREDIMED Study Investigators. Primary Prevention of Cardiovascular Disease with a Mediterranean Diet Supplemented with Extra-Virgin Olive Oil or Nuts. N Engl J Med. 2018 Jun 21;378(25):e34. doi: 10.1056/NEJMoa1800389. Epub 2018 Jun 13. PMID 29897866
- [Background] Wang DD, Li Y, Chiuve SE, Stampfer MJ, Manson JE, Rimm EB, Willett WC, Hu FB. Association of Specific Dietary Fats With Total and Cause-Specific Mortality. JAMA Intern Med. 2016 Aug 1;176(8):1134-45. doi: 10.1001/jamainternmed.2016.2417. PMID 27379574
- [Background] Wheeler ML, Dunbar SA, Jaacks LM, Karmally W, Mayer-Davis EJ, Wylie-Rosett J, Yancy WS Jr. Macronutrients, food groups, and eating patterns in the management of diabetes: a systematic review of the literature, 2010. Diabetes Care. 2012 Feb;35(2):434-45. doi: 10.2337/dc11-2216. No abstract available. PMID 22275443
- [Background] Brown TJ, Brainard J, Song F, Wang X, Abdelhamid A, Hooper L; PUFAH Group. Omega-3, omega-6, and total dietary polyunsaturated fat for prevention and treatment of type 2 diabetes mellitus: systematic review and meta-analysis of randomised controlled trials. BMJ. 2019 Aug 21;366:l4697. doi: 10.1136/bmj.l4697. PMID 31434641
- [Background] Arulselvan P, Fard MT, Tan WS, Gothai S, Fakurazi S, Norhaizan ME, Kumar SS. Role of Antioxidants and Natural Products in Inflammation. Oxid Med Cell Longev. 2016;2016:5276130. doi: 10.1155/2016/5276130. Epub 2016 Oct 10. PMID 27803762
- [Background] Kizil M, Tengilimoglu-Metin MM, Gumus D, Sevim S, Turkoglu I, Mandiroglu F. Dietary inflammatory index is associated with serum C-reactive protein and protein energy wasting in hemodialysis patients: A cross-sectional study. Nutr Res Pract. 2016 Aug;10(4):404-10. doi: 10.4162/nrp.2016.10.4.404. Epub 2016 Mar 29. PMID 27478547